CLINICAL TRIAL: NCT05623800
Title: HIV Education Kit for Adolescents (Pencegahan HIV di Kalangan Remaja), PREM-Kit
Acronym: PREM-Kit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Teknologi Mara (Other)
Responsible Party: Principal Investigator, Wan Nur Syamimi Binti Wan Mohamad Darani, Principal Investigator, Universiti Teknologi Mara
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REC/05/2022 (ST/MR/85)
Record Dates: First submitted 2022-11-03; First posted 2022-11-21 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Human Immunodeficiency Virus
Keywords: Human Immunodeficiency Virus; Adolescents; Information-Motivation-Behavioral Skills Model
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PREM-Kit group (Experimental)
  Interventions: Other: PREM-Kit
- Control group (No Intervention)

INTERVENTIONS:
Other: PREM-Kit — The PREM-Kit, which was created based on the Information-Motivation-Behavioral Skills model, is used in a series of HIV education sessions as part of the intervention. Over the course of three sessions, there will be a total of six weeks (one session for every two weeks). Three sub-modules, namely HIV facts and information, motivation for HIV preventive behavior, and behavioral skills for HIV prevention, will be emphasized in each session to the participants via flip chart and health educational videos. Additionally, participants will receive a QR code that gives them access to the PREM-Kit's e-flip chart, which they can see at a later time.
  Arms: PREM-Kit group

SUMMARY:
The goal of this community trial is to provide HIV education based on the newly developed HIV education kit (PREM-Kit) and evaluate the knowledge, attitude and practices related to HIV prevention among the late adolescents (aged 18 to 19 years old) in Malaysia. The main question it aims to answer is does the PREM-Kit improve the knowledge, attitude and practices related to HIV prevention among the adolescent?

Participants will be asked to:

* answer a questionnaire as a baseline screening to determine their knowledge, attitude and practices related to HIV prevention.
* Using PREM-Kit, they will participate in a series of health education sessions. There will be three sessions in total which will be delivered two weekly apart. Each of the sessions will take approximately 20 minutes duration.
* Following the last session (third session), participants will have to answer the same questionnaire ; once immediately after the last session, once at 3-months post-intervention, and lastly, at 4-months post-intervention.

Researchers will compare participants who received the existing Basic Science and Biology module to see if there is any improvement in the knowledge, attitude and practices related to HIV prevention.

ELIGIBILITY:
Inclusion Criteria:

* late adolescents aged 18 - 19 years
* student who attends Health Science Diploma course in the year 2023
* Malaysian citizen

Exclusion Criteria:

* student who refused to participate in the study
* student who is absent on the first session of the intervention
* student who does not understand the Malay language

Ages: 18 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 189 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-08-03 (Actual)

PRIMARY OUTCOMES:
Change in knowledge score related to HIV prevention | t1:Measurement of knowledge score before intervention. t2:Measurement of knowledge score immediately post-intervention. t3:Measurement of knowledge score at 3-months post-intervention. t4:Measurement of knowledge score at 4-months post-intervention.
  Knowledge score will be determined by using 15 questions related to HIV/AIDS transmission and prevention. The participants will be asked to respond on the individual statement using "Yes" or "No" or "I do not know" response. Each correct answer will be credited with 1 point, whereas wrong answers and ''I don't know'' answers will be assigned 0 points. The sum calculated to determine a total score for this scale. The possible range of total score is 0 to 15, where higher score indicates higher level of knowledge.
Change in attitude score related to HIV prevention | t1:Measurement of attitude score before intervention. t2:Measurement of attitude score immediately post-intervention. t3:Measurement of attitude score at 3-months post-intervention. t4:Measurement of attitude score at 4-months post-intervention.
  To assess the attitude score, eight items are used to assess the participants' attitude toward HIV/AIDS prevention. It consists of 5-point Likert scale (strongly agree, agree, undecided, disagree and strongly disagree). The scale given to the answers which is positive or agreeable is in the order of 5, 4, 3, 2, and 1. The scale given to the negative answers is in the reverse order. The possible range of the total score is 8 to 40, where higher score indicates higher positive attitude related to HIV prevention.
Change in practice score related to HIV prevention | t1:Measurement of practice score before intervention. t2:Measurement of practice score immediately post-intervention. t3:Measurement of practice score at 3-months post-intervention. t4:Measurement of practice score at 4-months post-intervention.
  Practice score will be assessed by six questions. All practice items are measured by "Yes", "No" and "I do not know" response. For questions such as (i) Do you watch any form of pornography?, (ii) Do you smoke?, (iii) Have you ever drink alcohol?, (iv) Have you ever tried any narcotic drugs?, and (v) Have you ever had sexual intercourse?, the "Yes" and "I do not know" responses will be scored as 0 point and "No" response will be scored as 1. On the other hand, the question of (vi) Have you ever talked about AIDS or HIV infection with your parents or other adults in your family?, "Yes" response will score 1 point, whereas, "No" and "I do not know" response will score 0. The possible range of total score of this practice measure is between 0 to 6, where higher score is indicative for more good practices related to HIV prevention.

CONTACTS AND LOCATIONS:
Overall Officials: Wan Nur Syamimi N Wan Mohamad Darani, Principal Investigator
Locations (2):
- Malaysia (2):
  - Universiti Teknologi MARA (UiTM Campus Tapah), Tapah, Perak
  - Universiti Teknologi MARA (Bertam Campus), Kepala Batas, Pulau Pinang

IPD SHARING:
Plan to Share IPD: No